CLINICAL TRIAL: NCT00890968
Title: A Multi-Center Randomized, Double-Blind, Placebo Controlled, Parallel Group Comparison Study of Once Daily Triamcinolone Acetonide 0.5% DuraPeel™ Versus Placebo DuraPeel in the Treatment of Hand Dermatitis
Brief Title: Safety and Efficacy Study of Triamcinolone Acetonide DuraPeel to Treat Hand Dermatitis
Acronym: TAC-202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAC-202
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Hand Dermatoses
Keywords: hand dermatitis; hand eczema; triamcinolone acetonide
MeSH Terms: conditions — Hand Dermatoses | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triamcinolone Acetonide (TAC) DuraPeel (Experimental)
  Interventions: Drug: Triamcinolone Acetonide (TAC) DuraPeel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo DuraPeel

INTERVENTIONS:
Drug: Triamcinolone Acetonide (TAC) DuraPeel — topical gel; once daily (nightly); total duration: 4 weeks
  Other Names: TAC DuraPeel
  Arms: Triamcinolone Acetonide (TAC) DuraPeel
Drug: Placebo DuraPeel — topical gel; once daily (nightly); total duration: 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Triamcinolone Acetonide (TAC) DuraPeel is safe and effective in the treatment of hand dermatitis.

DETAILED DESCRIPTION:
Triamcinolone acetonide is a commonly used, safe, and effective topical corticosteroid indicated for the relief of the inflammatory and pruritic manifestations of corticosteroid-responsive dermatoses. However, the effectiveness of topical agents such as creams or ointments is limited by patients' routine activities using bare hands that may remove the topical agent from the hands. The use of a topical corticosteroid in a vehicle that allows the product to remain in contact with the skin and is not susceptible to inadvertent removal would be beneficial.

The DuraPeel membrane is expected to optimize exposure to the steroid by remaining on the treatment area for a prolonged period of time.

This study is designed to evaluate the efficacy and safety of Triamcinolone Acetonide 0.5% DuraPeel. Eligible subjects will receive Triamcinolone Acetonide 0.5% DuraPeel or Placebo DuraPeel. The study duration will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stable chronic hand dermatitis (greater than 6 weeks duration) that is KOH-negative
* Dermatitis of mild to moderate severity, as defined by an Investigator's Global Assessment (a score of 2 or 3 on the Target Hand)
* Individual signs of hand dermatitis disease of at least mild scaling and mild erythema (a score of 2 or more on the Target Hand)
* Written informed consent

Exclusion Criteria:

* Subject is female and is pregnant, lactating, or is planning to become pregnant during the study
* Spontaneously improving or rapidly deteriorating hand dermatitis at the time of enrollment; subject may have history of waxing and waning disease in the past
* History of hand dermatitis that has been shown to be unresponsive to super potent (Group 1) topical steroids
* Concurrent flaring of inflammatory skin disease (e.g., atopic dermatitis or psoriasis) anywhere on the body outside the study areas
* Bullous disorders or hand, foot, and mouth disease (HFMD); however, subjects with dyshidrotic hand dermatitis or pompholyx are allowed to participate provided they meet all other Inclusion/Exclusion criteria
* Known allergic mediated hand dermatitis (e.g., allergic to latex, etc.)
* Concurrent skin diseases in the study area that require concomitant topical treatment (e.g., tinea manuum, scabies, infected eczema, and paronychia) that could interfere with the evaluation of his/her dermatitis
* Pustular diseases of the hands (e.g., acrodermatitis perstans continua).
* Used photo-therapy, photo-chemotherapy, systemic immunomodulatory therapy (such as systemic corticosteroids, methotrexate, retinoids or cyclosporine), or other therapy within 30 days prior to the first application of study medication that is known or suspected, in the opinion of the investigator, to have an effect on hand dermatitis
* Prolonged exposure to natural or artificial sources (e.g., UVB, UVA, etc.) of ultraviolet radiation within 30 days prior to the first application of study medication or is intending to have such exposure during the study
* Received intralesional therapy to the hands (e.g., corticosteroids) within 30 days prior to first application of study medication
* Treated with Grenz ray or soft x-ray therapy to the hands within 6 months of first application of study medication
* Treated with topical hand therapy (e.g., tar, topical corticosteroids, topical retinoids, topical antimicrobials, topical calcineurin inhibitors, Burrow's solution soaks) within 7 days prior to first application of study medication that is known or suspected to have an effect on hand dermatitis
* Received systemic antibiotics for infections of the hands within 7 days prior to the first application of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Response as assessed by Investigator Global Assessment (IGA) | Baseline, Week 1, Week 2, Week 4

SECONDARY OUTCOMES:
Subject's Global Impression of Change (SGIC) | Week 4 (end-of-treatment)
Individual Primary Parameters of Hand Dermatitis | Baseline, Week 1, Week 2, Week 4
Signs or symptoms of hand dermatitis | Baseline, Week 1, Week 2, Week 4
Subject's self-assessment of overall hand disease | Baseline, Week 4
Study medication assessment | Week 1, Week 2, Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Piacquadio, MD, Study Director — Therapeutics, Inc.
Locations (3):
- United States (3):
  - Therapeutics Clinical Research, San Diego, California
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - DermResearch Inc., Austin, Texas